CLINICAL TRIAL: NCT00117143
Title: An Open-label, Unit Dose-finding Study Evaluating the Safety and Efficacy of Amgen Megakaryopoiesis Protein 2 (AMG 531) in Thrombocytopenic Subjects With Immune Thrombocytopenic Purpura (ITP)
Brief Title: Amgen Megakaryopoiesis Protein 2 (AMG 531) in Thrombocytopenic Subjects With Immune Thrombocytopenic Purpura (ITP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20010218
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2019-11

CONDITIONS: Thrombocytopenic Purpura
Keywords: Immune Thrombocytopenic Purpura; Idiopathic Thrombocytopenic Purpura; ITP; Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic; Purpura, Thrombocytopenic, Idiopathic; Thrombocytopenia | interventions — romiplostim

ARMS (1):
- Romiplostim (Experimental): Participants will receive a maximum of 2 administrations of romiplostim by subcutaneous injection, the first on day 1 of the study and the second on day 15 or 22 depending on the participant's platelet count. Romiplostim doses to be tested were 30, 100, 300, and 500 μg.
  Interventions: Drug: Romiplostim

INTERVENTIONS:
Drug: Romiplostim — Administered subcutaneously on day 1 and on day 15 or 22 if the platelet count was ≤ 50 x 10⁹/L and not rising, peak platelet count was ≤ 450 x 10⁹/L and no serious adverse events related to treatment were observed.
  Other Names: AMG 531; NPLATE

SUMMARY:
The purpose of this study is to assess the safety and tolerability of AMG 531 (romiplostim), a novel thrombopoiesis-stimulating peptibody, and its effect on platelet counts in adults with immune thrombocytopenic purpura.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 3 months history of ITP, regardless of splenectomy status, and completion of at least 1 prior treatment for ITP
* 2 of 3 pretreatment platelet counts that were less than 30 x 10^9/L (if not currently on ITP therapy) or less than 50 x 10^9/L (if currently receiving corticosteroids for ITP therapy)
* Ability to give informed consent

Exclusion Criteria:

* Known history of arterial thrombosis, active malignancy, or bone marrow stem cell disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-12-02 (Actual); Primary Completion 2004-07-19 (Actual); Study Completion 2004-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Cines DB, Wasser J, Rodeghiero F, Chong BH, Steurer M, Provan D, Lyons R, Garcia-Chavez J, Carpenter N, Wang X, Eisen M. Safety and efficacy of romiplostim in splenectomized and nonsplenectomized patients with primary immune thrombocytopenia. Haematologica. 2017 Aug;102(8):1342-1351. doi: 10.3324/haematol.2016.161968. Epub 2017 Apr 14. PMID 28411254
- [Background] Newland A, Caulier MT, Kappers-Klunne M, Schipperus MR, Lefrere F, Zwaginga JJ, Christal J, Chen CF, Nichol JL. An open-label, unit dose-finding study of AMG 531, a novel thrombopoiesis-stimulating peptibody, in patients with immune thrombocytopenic purpura. Br J Haematol. 2006 Nov;135(4):547-53. doi: 10.1111/j.1365-2141.2006.06339.x. PMID 17061981
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: FDA-approved Drug Labeling — http://www.nplate.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter study conducted in 6 centers in France, the Netherlands, and the United Kingdom.
Pre-assignment Details: Participants were enrolled sequentially into one of four dose cohorts. When the platelet count of the first participant who received the 500 μg dose increased above 650 × 10⁹ cells/L following the first dose, this cohort was discontinued, and subsequent participants were assigned to the 300 μg cohort.
Groups:
- Romiplostim 30 µg: Participants received 30 µg romiplostim by subcutaneous injection on day 1 and a possible second dose on day 15 or 22 depending on the participant's platelet count.
- Romiplostim 100 µg: Participants received 100 µg romiplostim by subcutaneous injection on day 1 and a possible second dose on day 15 or 22 depending on the participant's platelet count.
- Romiplostim 300 µg: Participants received 300 µg romiplostim by subcutaneous injection on day 1 and a possible second dose on day 15 or 22 depending on the participant's platelet count.
- Romiplostim 500 µg: Participants received 500 µg romiplostim by subcutaneous injection on day 1 and a possible second dose on day 15 or 22 depending on the participant's platelet count.
Period: Overall Study
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Started | 4 | 4 | 7 | 1
Received First Dose | 4 | 4 | 7 | 1
Received Second Dose | 4 | 4 | 6 | 0
Completed | 4 | 4 | 7 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg | Total
Number analyzed (Participants) | 4 | 4 | 7 | 1 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.3 (14.9) | 37.8 (13.4) | 53.9 (20.4) | 45.0 | 50.9 (17.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 4 | 1 | 10
  Male | 1 | 2 | 3 | 0 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 6 | 1 | 15
  Black | 0 | 0 | 1 | 0 | 1
Platelet Count [Mean (Standard Deviation); unit: 10⁹cells/L] | 13.0 (6.10) | 16.5 (10.4) | 16.4 (7.77) | 28.8 | 16.3 (8.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Time Frame: From first dose through 8 weeks after last dose of study drug (11 weeks)
Population: Participants who received at least 1 dose of romiplostim
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants
  All adverse events | 4 | 4 | 7 | 1
  Serious adverse events | 0 | 0 | 3 | 1
  Treatment-related adverse events | 1 | 3 | 3 | 1
  Serious treatment-related adverse events | 0 | 0 | 1 | 1
  Discontinuations due to adverse events | 0 | 0 | 0 | 0
  Deaths | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Positive Anti-Romiplostim Antibodies
Description: The presence or development of antibodies to romiplostim and endogenous thrombopoietin was assessed using a neutralizing bioassay. Antibody analyses were conducted on study days 29 and at the end-of-study visit (day 78). The number of participants with positive antibody binding at any time during the study is reported.
Time Frame: Days 29 and 78
Population: Participants who received at least 1 dose of romiplostim
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants
  Anti-romiplostim antibodies | 0 | 0 | 0 | 0
  Anti-thrombopoietin antibodies | 0 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants Who Achieved a Targeted Therapeutic Platelet Response
Description: Targeted therapeutic platelet response was defined as a (single) platelet count that was double the baseline level and between 50 and 450 × 10⁹ cells/L.
  Platelet count data after the use of rescue medication were not included; participants with no platelet count data were considered non-responders.
Time Frame: Baseline and after first dose (days 3, 5, 8, 10, 12, 15, and days 17 and 19 for participants dosed on day 22) and after second dose (days 17, 19, and 22 for participants dosed on day 15, and days 24, 26, 29, 32, 36, 43, 50, 64, and 78 in all participants)
Population: Participants who received at least 1 dose of romiplostim.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants
  After First Dose | 1 | 4 | 4 | 0
  After Second Dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Second Dose | 1 | 3 | 3 |
  After Both Doses: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Both Doses | 1 | 3 | 3 |

4. Secondary Outcome: Number of Participants With an Increase in Platelet Count of ≥ 20 x 10⁹ Cells/L From Baseline
Description: Platelet count data after the use of rescue medication were not included; participants with no platelet count data were considered non-responders.
Time Frame: as for outcome 3
Population: Participants who received at least 1 dose of romiplostim.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants
  After First Dose | 2 | 4 | 5 | 1
  After Second Dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Second Dose | 1 | 3 | 4 |
  After Both Doses: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Both Doses | 1 | 3 | 3 |

5. Secondary Outcome: Number of Participants With Peak Platelet Counts of ≥ 100 x 10⁹ Cells/L
Description: as for outcome 4
Time Frame: After first dose (days 3, 5, 8, 10, 12, 15, and days 17 and 19 for participants dosed on day 22), and after second dose (days 17, 19, and 22 for participants dosed on day 15, and days 24, 26, 29, 32, 36, 43, 50, 64, and 78 for all participants)
Population: Participants who received at least 1 dose of romiplostim.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants
  After First Dose | 1 | 3 | 3 | 1
  After Second Dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Second Dose | 0 | 1 | 2 |
  After Both Doses: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Both Doses | 0 | 1 | 1 |

6. Secondary Outcome: Number of Participants With Peak Platelet Counts of ≥ 450 x 10⁹ Cells/L
Description: as for outcome 4
Time Frame: as for outcome 5
Population: Participants who received at least 1 dose of romiplostim.
Measure: Count of Participants; unit: Participants
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
Participants
  After First Dose | 0 | 0 | 1 | 1
  After Second Dose: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Second Dose | 0 | 0 | 0 |
  After Both Doses: number analyzed (Participants) | 4 | 4 | 6 | 0
  After Both Doses | 0 | 0 | 0 |

7. Secondary Outcome: Change From Baseline to Peak Platelet Level
Description: Platelet count data after the use of rescue medication were not included.
Time Frame: as for outcome 3
Population: Participants who received at least 1 dose of romiplostim with available data.
Measure: Mean (Standard Deviation); unit: 10⁹ cells/L
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
10⁹ cells/L
  After First Dose | 38.75 (50.50) | 89.98 (34.44) | 271.3 (558.4) | 1033.20 (NA) — Cannot be calculated for 1 participant
  After Second Dose: number analyzed (Participants) | 4 | 4 | 5 | 0
  After Second Dose | 11.50 (14.51) | 46.48 (25.15) | 56.38 (35.00) |

8. Secondary Outcome: Time to Peak Platelet Count
Description: Time from the date of study drug administration (day 1, 15 or 22) to the day of peak platelet count after each dose. Platelet count data after the use of rescue medication were not included.
Time Frame: From first dose of study drug to day 15 or 22, and from the second dose of study drug (day 15 or 22) to day 78
Population: Participants who received at least 1 dose of romiplostim with available data.
Measure: Median (Full Range); unit: days
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 4 | 4 | 7 | 1
days
  After First Dose | 10.5 [8 to 11] | 9.0 [5 to 10] | 12.0 [8 to 13] | 17.0 [17 to 17]
  After Second Dose: number analyzed (Participants) | 4 | 4 | 5 | 0
  After Second Dose | 13.5 [4 to 31] | 9.5 [8 to 12] | 9.0 [5 to 15] |

9. Secondary Outcome: Duration Within the Targeted Therapeutic Range
Description: Targeted therapeutic platelet level was defined as a platelet count that was double the baseline level and between 50 and 450 × 10⁹ cells/L.
  Platelet count data after the use of rescue medication were not included.
Time Frame: From first dose of study drug to day 15 or 22, and from the second dose of study drug (day 15 or 22) to day 78
Population: Participants who received at least 1 dose of romiplostim with a targeted therapeutic response.
Measure: Median (Full Range); unit: days
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Number analyzed (Participants) | 1 | 4 | 4 | 0
days
  After First Dose | 10.0 [10 to 10] | 5.5 [1 to 7] | 8.0 [5 to 15] |
  After Second Dose: number analyzed (Participants) | 1 | 3 | 3 | 0
  After Second Dose | 1.0 [1 to 1] | 2.0 [2 to 5] | 8.0 [1 to 49] |

ADVERSE EVENTS:
Time Frame: From first dose through 8 weeks after last dose of study drug (11 weeks).
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Romiplostim 30 µg | Romiplostim 100 µg | Romiplostim 300 µg | Romiplostim 500 µg
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 3/7 | 1/1
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 7/7 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim 30 µg (N=4) | Romiplostim 100 µg (N=4) | Romiplostim 300 µg (N=7) | Romiplostim 500 µg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim 30 µg (N=4) | Romiplostim 100 µg (N=4) | Romiplostim 300 µg (N=7) | Romiplostim 500 µg (N=1)
Thrombocythaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral mucosal petechiae (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 3 | 0
Injection site haemorrhage (General disorders) | 1 | 1 | 1 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 3 | 0
Ear infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Headache (Nervous system disorders) | 0 | 3 | 4 | 1
Lethargy (Nervous system disorders) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin bleeding (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1 | 1
Petechiae (Vascular disorders) | 0 | 2 | 1 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.